CLINICAL TRIAL: NCT04302142
Title: Effect of Applying Cuff Air Leak Pressure as Intraoperative Cuff Pressure on Postoperative Complications: Prospective Randomized Control Trial
Brief Title: Effect of Applying Cuff Air Leak Pressure as Intraoperative Cuff Pressure on Postoperative Complications
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to COVID restrictions on staff, therefore enrollment was not started.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Yandong Jiang, Visiting Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HSC-MS-20-0018
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Intubation Complication
Keywords: anesthesia; endotracheal tube cuff pressure
MeSH Terms: interventions — Polymerase Chain Reaction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Device: ventilation with critical intracuff pressure (Pcr)
- Control Group (Placebo Comparator)
  Interventions: Device: ventilation with critical intracuff pressure (Pcr)

INTERVENTIONS:
Device: ventilation with critical intracuff pressure (Pcr) — Once the intra-cuff pressure is measured and recorded, the cuff will be deflated by drawing the air 0.5ml per step with each step lasting 3 breaths until a leak, in which a 10% reduction in expiratory volume over the inspiratory tidal volume, is detected.Cuff will then be reinflated until the expiratory tidal volume reaches the inspiratory tidal volume and the discrepancy between the inspiratory and expiratory tidal volume is less than 10 percent. If the intra-cuff pressure applied by the anesthesia care team is inadequate and the discrepancy between the inspiratory and expiratory tidal volume is 10% or greater, the cuff will be further inflated with air 0.5ml per step with each step lasting 3 breaths until it reaches Pcr. This Pcr will be maintained during the entire anesthesia time until extubation.During the course of surgery, if any leak is detected, the cuff will be re-inflated by 0.5ml of air until the leak is not detectable.
  Arms: Intervention group
Device: ventilation with critical intracuff pressure (Pcr) — Pcr is obtained just as it is done in the intervention group. The cuff will then be reinsufflated to the actual cuff pressure the care team initially chose. The care team will be blinded to the measured critical cuff pressures and hence will maintain the usual level of intracuff pressure in the control group during the entire anesthesia time.
  Arms: Control Group

SUMMARY:
The purpose of the study is to achieve effective ventilation with critical intracuff pressure (Pcr) and determine if application of Pcr reduces the risks associated with over-insufflation of endotracheal cuff including postoperative sore throat, cough,nausea, vomiting, aspiration, and pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Elective Surgery under general anesthesia requiring endotracheal tube with mechanical ventilation and expected anesthesia duration of at least 2 hours.
* No contra-indication for intra-operative volume controlled mechanical ventilation
* Flat supine surgeries without expected positional adjustments
* American Society of Anesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* Use of Nitrous Oxide
* BMI > 40
* Ventilation through Nasal intubation or Tracheostomy
* Preexisting sore throat, coughing, nausea/vomiting
* Recent history of upper respiratory infection
* Pregnancy
* Expected to be kept intubated after surgery completion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Minimum intracuff pressure at which there is no air leak around the cuff. | during surgery

SECONDARY OUTCOMES:
Number of patients with postoperative sore throat as measured by a standardized questionnaire | 30 minutes post extubation
  The questionnaire utilizes a 4 point scale ,0 being mild and 3 being severe
Number of patients with postoperative sore throat as measured by a standardized questionnaire | 2 hours post extubation
  The questionnaire utilizes a 4 point scale ,0 being mild and 3 being severe
Number of patients with postoperative sore throat as measured by a standardized questionnaire | 24 hours post extubation
  The questionnaire utilizes a 4 point scale ,0 being mild and 3 being severe
Number of patients with postoperative coughing as measured by a standardized questionnaire | 30 minutes post extubation
  The questionnaire utilizes a 4 point scale ,0 being mild and 3 being severe
Number of patients with postoperative coughing as measured by a standardized questionnaire | 2 hours post extubation
  The questionnaire utilizes a 4 point scale ,0 being mild and 3 being severe
Number of patients with postoperative coughing as measured by a standardized questionnaire | 24 hours post extubation
  The questionnaire utilizes a 4 point scale ,0 being mild and 3 being severe
Number of patients with postoperative nausea/vomiting as measured by a standardized questionnaire | 30 minutes post extubation
  The questionnaire utilizes a 4 point scale ,0 being mild and 3 being severe
Number of patients with postoperative nausea/vomiting as measured by a standardized questionnaire | 2 hours post extubation
  The questionnaire utilizes a 4 point scale ,0 being mild and 3 being severe
Number of patients with postoperative nausea/vomiting as measured by a standardized questionnaire | 24 hours post extubation
  The questionnaire utilizes a 4 point scale ,0 being mild and 3 being severe
Number of patients with postoperative aspiration as measured by a standardized questionnaire | 30 minutes post extubation
  The questionnaire utilizes a 4 point scale ,0 being mild and 3 being severe
Number of patients with postoperative aspiration as measured by a standardized questionnaire | 2 hours post extubation
  The questionnaire utilizes a 4 point scale ,0 being mild and 3 being severe
Number of patients with postoperative aspiration as measured by a standardized questionnaire | 24 hours post extubation
  The questionnaire utilizes a 4 point scale ,0 being mild and 3 being severe

CONTACTS AND LOCATIONS:
Overall Officials: Yandong Jiang, MD,PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No